CLINICAL TRIAL: NCT00324350
Title: Intensive Glycemic Control and Skeletal Health Study - Ancillary Study to the Action to Control Cardiovascular Risk in Diabetes Trial (ACCORD-BONE)
Brief Title: Intensive Glycemic Control and Skeletal Health Study
Acronym: ACCORD-BONE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: R01DK069514 (NIH)
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-09

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Hypercholesterolemia; Hypertension; Diabetes Mellitus; Coronary Disease
Keywords: Diabetes Mellitus; Fracture; Falls; Height Loss
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Hypercholesterolemia; Hypertension; Diabetes Mellitus; Coronary Disease; Fractures, Bone | interventions — Hypoglycemic Agents; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): intensive glycemic control (therapeutic strategy that targets a glycosylated hemoglobin (HbA1c) level below 6.0%)
  Interventions: Drug: hypoglycemic agents, hydroxymethylglutaryl-CoA Reductase inhibitors, hypertensive agents
- 2 (Active Comparator): standard glycemic control (therapeutic strategy that targets a glycosylated hemoglobin (HbA1c) level of 7 to 7.9%)
  Interventions: Drug: hypoglycemic agents, hydroxymethylglutaryl-CoA Reductase inhibitors, hypertensive agents

INTERVENTIONS:
Drug: hypoglycemic agents, hydroxymethylglutaryl-CoA Reductase inhibitors, hypertensive agents — type 2 diabetes treatments, per standard of care

SUMMARY:
The purpose of the ACCORD-BONE Study is to investigate the effects of intensive glycemic control for type 2 diabetes (in ACCORD participants) on factors related to bone health, including, fractures, falls, and bone mineral density.

DETAILED DESCRIPTION:
Recent studies have established that type 2 diabetes is a risk factor for fractures, particularly of the hip, shoulder and foot. Additionally, type 2 diabetes is associated with a 50-60% increase in the risk of falling. The higher risk of fracture associated with type 2 diabetes is an important health burden for these patients. More frequent falls and perhaps reduced bone strength in those with diabetes are thought to be key contributing factors. The best approach to preventing fractures in type 2 diabetes is not yet understood. There is observational evidence to support our hypothesis that better glycemic control will preserve bone and reduce falls and fractures. The ACCORD-BONE study provides a unique opportunity to determine whether intensive glycemic control will prevent fractures, falls, and bone loss in older diabetic adults, which may lead to improved treatment and prevention in the future.

ELIGIBILITY:
Inclusion criteria:

* Fulfills criteria for inclusion in the ACCORD main trial
* Must have been randomized into the ACCORD study and be a participant from the five CCNs in the ACCORD-BONE ancillary study.

Exclusion criteria:

* Fulfills criteria for exclusion in the ACCORD main trial

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7287 (Actual)
Dates: Start 2003-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann V. Schwartz, PhD, Principal Investigator — University of California, San Francisco
Locations (5):
- United States (4):
  - Berman Center for Outcomes & Clinical Research, Minneapolis, Minnesota
  - Wake Forest University, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Veterans Affairs, Memphis, Tennessee
- Population Health Research Institute, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Schwartz AV, Margolis KL, Sellmeyer DE, Vittinghoff E, Ambrosius WT, Bonds DE, Josse RG, Schnall AM, Simmons DL, Hue TF, Palermo L, Hamilton BP, Green JB, Atkinson HH, O'Connor PJ, Force RW, Bauer DC. Intensive glycemic control is not associated with fractures or falls in the ACCORD randomized trial. Diabetes Care. 2012 Jul;35(7):1525-31. doi: 10.2337/dc11-2184. PMID 22723583
- [Derived] Schwartz AV, Chen H, Ambrosius WT, Sood A, Josse RG, Bonds DE, Schnall AM, Vittinghoff E, Bauer DC, Banerji MA, Cohen RM, Hamilton BP, Isakova T, Sellmeyer DE, Simmons DL, Shibli-Rahhal A, Williamson JD, Margolis KL. Effects of TZD Use and Discontinuation on Fracture Rates in ACCORD Bone Study. J Clin Endocrinol Metab. 2015 Nov;100(11):4059-66. doi: 10.1210/jc.2015-1215. Epub 2015 Aug 25. PMID 26305617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The ACCORD trial has been described previously (Buse JB,et al. Am J Cardiol 99:21i-33i, 2007). Five of the 7 clinical center networks agreed to participate in the BONE ancillary study, including 54 of 77 clinical sites and 7,287 participants. The BONE ancillary study was initiated during the main recruitment for ACCORD (beginning in 2006).
Groups:
- Intensive Glycemic Control: intensive therapeutic strategy targeting normal glycated hemoglobin (A1C) levels (i.e., below 6.0%)in a population with long-standing type 2 diabetes and a history of cardiovascular disease or significant cardiovascular risk factors
- Standard Glycemic Control: standard strategy targeting A1C levels from 7.0 to 7.9% in a population with long-standing type 2 diabetes and a history of cardiovascular disease or significant cardiovascular risk factors
Period: Overall Study
Arm/Group | Intensive Glycemic Control | Standard Glycemic Control
Started | 3655 | 3632
Non-Vertebral Fracture Follow-Up | 3655 | 3632
Falls Follow-Up | 3364 | 3418
Completed | 3655 | 3632
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Glycemic Control | Standard Glycemic Control | Total
Number analyzed (Participants) | 3655 | 3632 | 7287
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2380 | 2361 | 4741
  >=65 years | 1275 | 1271 | 2546
Age Continuous [Mean (Standard Deviation); unit: years] | 62.5 (6.7) | 62.6 (6.7) | 62.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1267 | 1251 | 2518
  Male | 2388 | 2381 | 4769
Region of Enrollment [Number; unit: participants]
  United States | 2903 | 2876 | 5779
  Canada | 752 | 756 | 1508

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Non-vertebral Fracture
Description: The BONE ancillary study was initiated during recruitment for the main ACCORD trial. Beginning in January 2006, at the next annual visit participants were asked about the occurrence of any non-spine fractures since randomization. After the annual visit in 2006, participants were asked if they had suffered a fracture since their last annual visit. Reported fracture events were centrally adjudicated, based on radiology records, at the University of California, San Francisco (UCSF) with the adjudicators blinded to treatment assignment.
Time Frame: Average follow-up of 3.8 years
Population: As per protocol, pathological fractures, confirmed as occurring secondary to neoplasm, necrosis, or sepsis, and periprosthetic fractures were excluded (N=7). These analyses are limited to confirmed fractures that occurred on or before Feb 5, 2008, when the intensive glycemia intervention was ended.
Measure: Number; unit: participants
Arm/Group | Intensive Glycemic Control | Standard Glycemic Control
Number analyzed (Participants) | 3655 | 3632
participants | 198 [.86 to .127] | 189
Statistical Analysis 1: Comparison: Intensive Glycemic Control vs Standard Glycemic Control; The BONE ancillary study was designed to have 80% power to detect a relative reduction in risk of non-spine clinical fractures of 22-29%. This was based on an estimated total number of fractures between 259-494, calculated with the following assumptions: rate of clinical non-spine fracture among women in the standard glycemia therapy group between 15 and 25/1000 person yrs, fracture rates for men between 35-40% of the rates for women of the same age, and an avg follow-up time of 4.6 yrs; Test type: Superiority or Other; p = 0.678, Regression, Cox — Analyses were by intention to treat. All analyses adjusted for baseline cardiovascular disease, assignment to blood pressure (BP) trial or lipid trial, assignment to intensive BP intervention in BP trial, and assignment to fibrate in lipid trial; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.86 to 1.27]

2. Primary Outcome: Number of Participants With at Least One Fall
Description: At each annual visit starting in January 2006, participants were also asked about falling: "In the last 12 months have you fallen and landed on the floor or ground, OR fallen and hit an object like a table or stair?" Those who answered "yes" were also asked how many times they had fallen in the previous 12 months.
Time Frame: Average follow-up of 2.0 years
Population: These analyses include results from the annual visits that occurred before Feb 5, 2008, the close of the intensive glycemia arm. Of those in the BONE ancillary study, 6,782 participants answered at least one question about falls.
Measure: Number; unit: participants
Groups:
- Intensive Glycemic Control: intensive therapeutic strategy targeting normal glycated hemoglobin (A1C) levels (i.e., below 6.0%) in a population with long-standing type 2 diabetes and a history of cardiovascular disease or significant cardiovascular risk factors
Arm/Group | Intensive Glycemic Control | Standard Glycemic Control
Number analyzed (Participants) | 3364 | 3418
participants | 1122 | 1133
Statistical Analysis 1: Comparison: Intensive Glycemic Control vs Standard Glycemic Control; Number of participants with falls reported at each annual visit were compared by treatment assignment using a repeated-measures negative binomial model, with robust standard errors to account for clustering of the repeated outcomes within participants; the log of the length of the reporting period varied slightly and was included as an offset; Test type: Superiority or Other; p = 0.490, Regression, Cox; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.84 to 1.43]

3. Secondary Outcome: Number of Participants With > 2 cm of Height Loss
Description: Standing height was measured according to a standard protocol at baseline and annual visits on all ACCORD participants. Height loss was compared by treatment assignment using linear mixed models with random intercepts and slopes. Treatment effects were captured by the interaction between treatment assignment and time. The proportions losing >2 cm of height during follow-up were compared using logistic models. This degree of height loss is associated with incident vertebral fracture with 94% specificity but only 28% sensitivity
Time Frame: 5 years
Population: Among participants in the BONE ancillary study, 6,979 participants had at least one height measurement during follow-up and were included in these analyses.
Measure: Number; unit: participants
Arm/Group | Intensive Glycemic Control | Standard Glycemic Control
Number analyzed (Participants) | 3482 | 3497
participants | 678 | 686
Statistical Analysis 1: Comparison: Intensive Glycemic Control vs Standard Glycemic Control; Height loss was compared by treatment assignment using linear mixed models with random intercepts and slopes. The proportions losing >2 cm of height during follow-up were compared using logistic models. Based on previous research by Siminoski et al., this degree of height loss is associated with incident vertebral fracture with 94% specificity but only 28% sensitivity.(Siminoski K, Jiang G, Adachi JD, et al. Osteoporos Int 2005;16:403-410); Test type: Superiority or Other; p = 0.854, Mixed Models Analysis; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.88 to 1.11] — The rate of height loss did not differ between groups (p = 0.573). Height loss of >2 cm during ACCORD was experienced by 678 (19.5%) participants in the intensive and 686 (19.6%) in the standard glycemia group (OR 0.99; 95% CI 0.88, 1.11)

ADVERSE EVENTS:
Description: Adverse events were not collected as a part of this ACCORD-BONE ancillary study. Please refer to the ACCORD main study results for all adverse event results.
Arm/Group | Intensive Glycemic Control | Standard Glycemic Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The initial identification of a possible fracture event relied on self-report at annual visits with the possibility of under- or over-reporting of fractures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No